CLINICAL TRIAL: NCT05421949
Title: Assessing the Repeatability of NT-proBNP Testing Using Laboratory and Point of Care Testing in PAH (REPEAT-PAH)
Brief Title: Assessing the Repeatability of NT-proBNP Testing Using Laboratory and Point of Care Testing in PAH
Acronym: REPEAT-PAH
Status: Completed | Type: Observational
Sponsor: Sheffield Teaching Hospitals NHS Foundation Trust (Other)
Collaborators: Actelion (Industry)
Responsible Party: Sponsor
Other Study IDs: STH20981
Record Dates: First submitted 2022-06-07; First posted 2022-06-16 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Pulmonary Artery Hypertension
MeSH Terms: conditions — Familial Primary Pulmonary Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Exercise: Patients who have been randomised to the exercise group will be asked to undertake a incremental shuttle walking test following their initial blood tests.
  Interventions: Other: Exercise group
- No Exercise: Patients who have been randomised to the exercise group will be asked to rest for 60 minutes following their initial blood tests.

INTERVENTIONS:
Other: Exercise group — Incremental Shuttle Walking Test
  Groups: Exercise

SUMMARY:
The purpose of this study is to examine N-terminal pro brain natriuretic peptide (NT-proBNP) and brain natriuretic peptide (BNP) biomarkers in a number of different settings including assessing the repeatability of laboratory and point of care testing (POCT), the effect of a time delay and exercise have on laboratory measurements. Also to compare the clinical and analytical performances of NT-proBNP and BNP POCT samples across the spectrum of disease severity and finally assess whether POCT in PAH can detect change in patients commencing or escalating PAH treatment.

DETAILED DESCRIPTION:
* Patients that are attending clinical appointments will be approached to ask if they will take part in the study.
* Patients will be assessed at two separate visits.
* Patients will be randomised to either exercise or rest group on their 1st visit. On the 2nd visit patients will be asked to participate in the alternate group to what they completed on their previous visit.
* At each visit they will have 2 blood samples taken, at time point 1 and at time point 2 (T1 and T2). These will be taken at least one hour apart, each with a period of at least 15 mins rest in the sitting position prior to sampling.
* On one of these two visits the patient will undergo exercise testing between T1 and T2.
* In addition, a further laboratory testing tube will be taken for a delayed NT-proBNP. This will be subjected to gentle agitation (laboratory rotator) for 48 hours prior to processing to simulate, in a controlled environment, the effect of transport and delay on sample measurement.
* Retrospectively information will be collected regarding the patient's disease severity and any change to treatment that occurred between the two visits.
* A total of 40 patients with be sampled with an interim analysis after 20 patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have met the criteria for The Sheffield Teaching Hospitals Observational Study of Patients with Pulmonary Hypertension, Cardiovascular and other Respiratory Diseases (STH-ObS)
* Patient diagnosed with Group 1 PAH, including IPAH, HPAH, PAH-CTD but excluding PAH-CHD. Mean pulmonary artery pressure >20mmHg, PAWP ≤15mmHg and PVR >240 dynes.
* Willing to participate in the study and able to provide informed consent

Exclusion Criteria:

* Diagnosed with PAH-CHD or any non-group 1 PH
* Creatinine clearance < 15 ml/min/m2

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with pulmonary arterial hypertension
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2021-02-19 (Actual); Primary Completion 2022-08-30 (Actual); Study Completion 2022-08-30 (Actual)

PRIMARY OUTCOMES:
The repeatability of laboratory and POCT samples for NT-proBNP and BNP in patients at rest with PAH. | 18 months
  Comparisons will be made between time point 1 (T1) and 2 (T2) in the absence of exercise for venous blood using POCT kits and for venous blood using laboratory analysis, for both BNP and NT-proBNP.
The effect of a pre-processing time delay on performance of NT-proBNP test | 18 months
  Comparison will be made between samples sent directly to the laboratory and those that were delayed in being sent by 48 hours. Pre-specified levels will be used to determine the performance of the test as excellent (eg >=0.75), good, fair or poor.
The impact of exercise testing using the incremental shuttle walking test (ISWT) on NT-proBNP and BNP on both laboratory and POCT samples | 18 months
  Comparison will be made between venous blood using POCT kits and venous blood using laboratory testing at rest and post exercise, for both BNP and NT-proBNP.
The impact of treatment change or escalation on the results of POCT and The change in POCT and laboratory samples for NT-proBNP and BNP. | 18 months
  POCT and laboratory samples for NT-proBNP and BNP will be assessed to see if they detected change in patients who had a change or escalation in treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Pulmonary Vascular Disease Unit, Royal Hallamshire Hospital, Sheffield, South Yorkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Durrington C, Battersby C, Holt L, Fairman A, Strickland S, Salisbury T, Turton HA, Watson L, Smith I, Roman S, Ablott J, Hitchcock F, Roddis C, Oakes E, Wilshaw H, Woodrow I, Armstrong I, Charalampopoulos A, Elliot CA, Hameed A, Hamilton N, Hurdman JA, Lawrie A, Middleton JT, Zafar H, Rothman AMK, Condliffe R, Lewis RA, Kiely DG, Thompson AAR. NT-proBNP and BNP Testing in Pulmonary Arterial Hypertension: Point-of-Care and Remote Monitoring. Respirology. 2025 Nov;30(11):1094-1103. doi: 10.1111/resp.70087. Epub 2025 Jul 3. PMID 40611611